CLINICAL TRIAL: NCT06574750
Title: New HA Filler Versus Juvederm for Nasolabial Fold Correction
Brief Title: Effect of a New HA Filler in Correcting Nasolabial Fold
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Bo Ri Kim, Assistant professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-2105/684-001
Record Dates: First submitted 2024-08-22; First posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Aging Problems
MeSH Terms: interventions — Long-Term Synaptic Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- New HA filler (Curea) (Experimental): The left/right assignment was sealed in a nontransparent envelop.
  Interventions: Drug: CUREAⓇ (ARIBIO, Ltd., Seoul, Republic of Korea)
- Juvederm (Active Comparator): The left/right assignment was sealed in a nontransparent envelop.
  Interventions: Drug: JuvedermⓇ (Q-Med AB, Uppsala, Sweden)

INTERVENTIONS:
Drug: CUREAⓇ (ARIBIO, Ltd., Seoul, Republic of Korea) — Hyaluronic acid filler injection were administered into the mid-dermis of the nasolabial fold.
  Other Names: experimental group
  Arms: New HA filler (Curea)
Drug: JuvedermⓇ (Q-Med AB, Uppsala, Sweden) — Hyaluronic acid filler injection were administered into the mid-dermis of the nasolabial fold.
  Other Names: active control group
  Arms: Juvederm

SUMMARY:
The investigators aimed to evaluate the efficacy and safety of new HA filler for nasolabial fold correction

DETAILED DESCRIPTION:
A 24-week prospective, single-center, assessor-blinded, randomized, split-face study was conducted to compare the clinical efficacy and safety of new HA filler versus Juvederm for nasolabial fold correction

ELIGIBILITY:
Inclusion Criteria:

* Patients who had prominent NLFs with a WSRS score of 3 or 4 on both sides

Exclusion Criteria:

* patients with active facial skin diseases or history of severe allergies, autoimmune disorders, or hypersensitivity to HA or any of the excipients contained in the investigational filler
* participants who had used a local topical preparation (steroid and retinoid) within 2 weeks before the study
* participants who had undergone chemical peeling, laser procedures, or acne treatments within 4 months before the study
* participants who had been injected with other biomaterials, including HA within 6 months before the study.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2021-10-16 (Actual); Primary Completion 2023-05-08 (Actual); Study Completion 2023-05-08 (Actual)

PRIMARY OUTCOMES:
WSRS | at 24 weeks after treatment
  Wrinkle Severity Rating Scale from 1 (no visible fold) to 5 (extremely deep and long folds)

SECONDARY OUTCOMES:
GAIS | at 24 weeks after treatment
  Global Aesthetic Improvement Scale from 3 (very much improved) to -1 (worse).
Adverse events related to the procedure | up to 24 weeks
  Patients were required to report any adverse events up to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bo Ri Kim, M.D., Ph.D., Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim BR, Shin JW, Kim DW, Choung JJ, Jang Y, Lee SH, Seo BS, Huh CH. Efficacy and Safety of New Hyaluronic Acid Filler for Nasolabial Fold Correction: A Double-Blind, Randomized Trial. Plast Reconstr Surg. 2026 Feb 1;157(2):249-256. doi: 10.1097/PRS.0000000000012320. Epub 2025 Jul 21. PMID 40707029